CLINICAL TRIAL: NCT04764331
Title: A Pilot Study of Revian Red All LED Cap as a Novel Treatment for Central Centrifugal Cicatricial Alopecia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00071484
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Central Centrifugal Cicatricial Alopecia

STUDY DESIGN:
Intervention Model Description: 5 subjects who are willing to participate in a novel treatment for Revian Red All LED cap will be enrolled in this study. The cap uses two wavelengths of light, 620 nm and 660 nm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Other): Caps will be provided for each subjects will use the cap once daily for10-minute treatment regimen
  Interventions: Device: Revian Red All LED cap

INTERVENTIONS:
Device: Revian Red All LED cap — Cap that uses two wavelengths of light, 620 nm and 660 nm will be used once a day for 10 minutes.for treatment
  Other Names: Revian Red

SUMMARY:
Central centrifugal cicatricial alopecia (CCCA) is form of scarring hair loss that predominately affects middle-aged women of African descent.1 . Clinically, the natural progression of CCCA starts at the crown as roughly circular scarred patches, which evolve into scarred areas increasing in size circumferentially. Characteristically, the scar is often smooth and shiny, and the hair density in the affected area is frequently decreased. The hair remaining in the scarred areas is more brittle and shorter than the hair in unaffected areas. Since CCCA is a scarring disorder, it can cause permanent hair loss, dyesthesias, and psychological distress which can affect overall quality of life. Affected individuals may complain of pruritus, pain, or tenderness.2

The management of CCCA is challenging due to limited current treatments and a lack of randomized controlled trails. Management focuses on behavioral and styling modifications, in addition to symptomatic relief. Any potentially damaging hair care practices such as chemical relaxers, heat application to the scalp, and the use of hardening gels and sprays are discouraged.3 Many commonly used therapies are anti-inflammatory in nature, including intralesional steroids, topical steroids, oral antibiotics and increased frequency of hair washing with antidandruff shampoos.4 These treatments not only lead to improvement in pruritus and tenderness, but in some cases result in increased hair density.5 Since there is limited investigation done to determine the most effective treatment approach for CCCA subjects, it would be of great benefit to determine if there is any advantage in using one particular anti-inflammatory therapy over others and whether one is more efficacious in relieving symptoms or promoting hair regrowth in follicles that have not yet become scarred.

The Revian Red All LED cap is a dual-band LED light therapy wireless "smart" cap. It has been effective in androgenetic alopecia (used once daily, 10-minute treatment regimen) for both men and women. There are also reportedly minimal side effects, unlike with topical minoxidil which can cause pruritus and initial hair shedding in the first few weeks, or finasteride which can cause gynecomastia and loss of libido. In this study we hope to see if the anti-inflammatory capabilities of this cap can improve scalp symptoms, reduce hair loss, and promote maturation of vellus and intermediate hairs in non-scarred areas of the scalp in those affected by CCCA.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine if the Revian Red All LED cap shows potential to be an effective treatment for CCCA by recruiting hair follicles back to anagen growth or by improving inflammation. The primary outcome is to determine if hair loss regression is halted. Secondary outcomes include hair regrowth and alleviation of signs and symptoms of the disease.

Methods and Measures

Design 5 subjects who are willing to participate in a novel treatment for Revian Red All LED cap will be enrolled in this study. The cap uses two wavelengths of light, 620 nm and 660 nm. A study caps will be provided for each subject. Subjects will use the cap once daily, 10-minute treatment regimen which is the current androgenetic alopecia recommendation. The subjects will use the cap for a total of 6 months.

Standardized photos and dermatoscope photos before starting treatment and every 2 months for x 6 total months will be taken to assess hairline stabilization and potential for regrowth.

Prior to study enrollment, all participants will receive a detailed explanation of the purpose of the study and will undergo written informed consent. Clinical history of hair loss and history of prior treatment will be obtained by administering a standardized questionnaire to all subjects. Subjects will also fill out a questionnaire regarding symptoms of their hair loss at each subsequent treatment visit and at follow-up. In order to be eligible, subjects must be diagnosed clinically and histologically with CCCA. Diagnosis will be made only by a board-certified dermatologist.

ELIGIBILITY:
Inclusion Criteria:

* Women who are eighteen years of age or older with a biopsy-proven diagnosis of CCCA Stage II-III. They also must be on stable treatment without changes (on doxycycline, topical steroids, minoxidil and/or post 8 rounds of intralesional steroids) for at least 3 months.
* Subjects will be recruited from outpatient dermatology clinics at the Wake Forest Baptist Health Department of Dermatology.

Exclusion Criteria

* Subjects with other forms of hair loss that is not CCCA
* Prior treatment with light source for alopecia
* Males are excluded from this study since the prevalence of CCCA in males is so significantly low that it is difficult to find cases in a clinical setting

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
hairline stabilization | Change from baseline to month 2
  Pre treatment photographs will also be assessed to determine if further scalp hairline recession is present and to look for hair regrowth
hairline stabilization | Change from month 2 to month 4
  Post-treatment photographs will also be assessed to determine if further scalp hairline recession is present and to look for hair regrowth
hairline stabilization | Change from month 4 to month 6 (end of study)
  Post-treatment photographs will also be assessed to determine if further scalp hairline recession is present and to look for hair regrowth
hairline regrowth | Change from baseline to month 2
  Pre treatment photographs will be assessed to determine if further scalp hairline recession is present and to look for hair regrowth
hairline regrowth | Change from month 2 to month 4
  Post-treatment photographs will also be assessed to determine if further scalp hairline recession is present and to look for hair regrowth
hairline regrowth | Change from month 4 to month 6 (end of study)
  Post-treatment photographs will also be assessed to determine if further scalp hairline recession is present and to look for hair regrowth

SECONDARY OUTCOMES:
patient assessment of stabilization | baseline
  Questionnaire will be completed at baseline
patient assessment of stabilization | month 6
  Questionnaire will be completed at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Amy McMichael, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine - Dermatology Clinic, Winston-Salem, North Carolina, United States